CLINICAL TRIAL: NCT04305548
Title: Phase II Study on Trabectedin in Advanced Rearranged Mesenchymal Chondrosarcoma
Brief Title: Study on Trabectedin in Advanced Rearranged Mesenchymal Chondrosarcoma
Acronym: ISG-MCS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISG-MCS
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Mesenchymal Chondrosarcoma
MeSH Terms: conditions — Chondrosarcoma, Mesenchymal | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trabectedin (Experimental): Trabectedin: 1.5 mg/m² - 1.3 mg/m² (at investigator's discretion, with a top-dose of 2.6 total mg per cycle), given in 24-hour continuous infusion
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin — Treatment with trabectedin: 1.5 mg/m² - 1.3 mg/m² (at investigator's discretion, with a top-dose of 2.6 total mg per cycle), given in 24-hour continuous infusion

SUMMARY:
Prospective, uncontrolled, investigator-initiated, phase II clinical study to explore the activity of trabectedin in a population of patients aged ≥16 years with progressive, advanced (locally advanced or metastatic)

DETAILED DESCRIPTION:
Prospective, uncontrolled, multicenter, Italian, investigator-initiated, phase II clinical study to explore the activity of trabectedin in a population of patients aged ≥16 years with progressive, advanced (locally advanced or metastatic), HEY1-NCOA2 positive MCS) , pre-treated with anthracycline-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years old
2. Histological centrally confirmed diagnosis of skeletal or extra-skeletal MCS with the documented presence of HEY1-NCOA2 fusion
3. Locally advanced disease and/or metastatic disease
4. Measurable or evaluable disease with RECIST v1.1
5. Evidence of progression by RECIST v1.1 during the 6 months before study entry
6. Patients must be pre-treated with at least one prior chemotherapy treatment containing anthracyclines for the advanced phase of disease and with a maximum of 3 lines
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
8. Adequate bone marrow function
9. Adequate organ function
10. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation each cycle of chemotherapy.
11. Cardiac ejection fraction ≥50% as measured by echocardiogram
12. No history of arterial and/or venous thromboembolic event within the previous 12 months
13. The patient or legal representative must be able to read and understand the informed consent form and must have been willing to give written informed consent and any locally required authorisation before any study-specific procedures, including screening evaluations, sampling, and analyses.
14. Any other factors, that, at judgment of investigator, could affect the safety of the patients according to the available trabectedin safety data

Exclusion Criteria:

1. Other primary malignancy with <5 years clinically assessed disease free interval, except basal cell skin cancer, cervical carcinoma in situ or other neoplasm judged to entail a low risk of relapse
2. Previous treatment with radiation therapy within 14 days of first day of study drug dosing, or patients who have not recovered from adverse events due to agents previously administered
3. Previous radiotherapy to 25% of the bone marrow
4. Major surgery within 2 weeks prior to study entry
5. Participation in another clinical study with an investigational product, which last dose was taken less than 4 weeks prior to the start of the treatment.
6. Persistent toxicities (≥ grade 2) with the exception of alopecia, caused by previous anticancer therapies.
7. Pregnancy or breast feeding
8. Grade III/IV cardiac problems as defined by the New York Heart Association Criteria
9. Medical history of arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), or pulmonary embolism within 6 months prior to the initiation of study treatment
10. Known brain metastasis
11. Known chronic liver disease (i.e. chronic active hepatitis and cirrhosis)
12. Known diagnosis oh human deficiency virus (HIV) infection
13. Active or chronic hepatitis B or C requiring treatment with antiviral therapy
14. Medical history of hemorrhage or a bleeding event ≥ Grade 3 within 4 weeks prior to the initiation of study treatment
15. Evidence of any other serious or unstable illness, or medical, psychological, or social condition, that could jeopardize the safety of the subject and/or his/her compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results
16. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs
17. Expected non-compliance to medical regimens

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall tumour Response Rate, according to RECIST v 1. | At weeks 6
  Response rate according Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Choi criteria response rate | At weeks 6, 12,18, 30, 42
  Response rate according Choi criteria
Overall Survival | At 3 and 5 years
  Proportion of patients who are still alive at 36 and 60 months after have started the treatment
Progression Free Survival (PFS) | At 3 and 5 years
  Survival without disease progression
Clinical Benefit Rate | Month 6
  Proportion of patient alive, without disease progression, after 6 months of treatment.
Duration of response | At weeks 6, 12,18, 30, 42
  Duration of time between the date of first documented response and the date of first documented progression or death due to any cause
Adverse events related to the treatment | Week 3, week 6, week 9, week 12, week 18, week 24, week 36, week 48, week 60, week 72
  Safety in term of grading of adverse event is evaluate from the first treatment dose throughout the study according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Stacchiotti, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (7):
- Italy (7):
  - Nuovo Ospedale di Prato, Prato, Firenze
  - Policlinico Universitario Campus Biomedico, Roma, RM
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Istituto Ortopedico Rizzoli - Unit of Chemotherapy of Muscoloskeletal Tumors, Bologna
  - Fondazione IRCSS Istituto Nazionale dei Tumori, Milan
  - Ospedale Giaccone, Palermo
  - Istituti Fisioterapici Ospitalieri - Ospedale Regina Elena, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee AF, Hayes MM, Lebrun D, Espinosa I, Nielsen GP, Rosenberg AE, Lee CH. FLI-1 distinguishes Ewing sarcoma from small cell osteosarcoma and mesenchymal chondrosarcoma. Appl Immunohistochem Mol Morphol. 2011 May;19(3):233-8. doi: 10.1097/PAI.0b013e3181fd6697. PMID 21084965
- [Background] Wang L, Motoi T, Khanin R, Olshen A, Mertens F, Bridge J, Dal Cin P, Antonescu CR, Singer S, Hameed M, Bovee JV, Hogendoorn PC, Socci N, Ladanyi M. Identification of a novel, recurrent HEY1-NCOA2 fusion in mesenchymal chondrosarcoma based on a genome-wide screen of exon-level expression data. Genes Chromosomes Cancer. 2012 Feb;51(2):127-39. doi: 10.1002/gcc.20937. Epub 2011 Oct 27. PMID 22034177
- [Background] Morioka H, Takahashi S, Araki N, Sugiura H, Ueda T, Takahashi M, Yonemoto T, Hiraga H, Hiruma T, Kunisada T, Matsumine A, Susa M, Nakayama R, Nishimoto K, Kikuta K, Horiuchi K, Kawai A. Results of sub-analysis of a phase 2 study on trabectedin treatment for extraskeletal myxoid chondrosarcoma and mesenchymal chondrosarcoma. BMC Cancer. 2016 Jul 14;16:479. doi: 10.1186/s12885-016-2511-y. PMID 27418251
- [Background] Forni C, Minuzzo M, Virdis E, Tamborini E, Simone M, Tavecchio M, Erba E, Grosso F, Gronchi A, Aman P, Casali P, D'Incalci M, Pilotti S, Mantovani R. Trabectedin (ET-743) promotes differentiation in myxoid liposarcoma tumors. Mol Cancer Ther. 2009 Feb;8(2):449-57. doi: 10.1158/1535-7163.MCT-08-0848. Epub 2009 Feb 3. PMID 19190116
- [Background] Huvos AG, Rosen G, Dabska M, Marcove RC. Mesenchymal chondrosarcoma. A clinicopathologic analysis of 35 patients with emphasis on treatment. Cancer. 1983 Apr 1;51(7):1230-7. doi: 10.1002/1097-0142(19830401)51:73.0.co;2-q. PMID 6825046